CLINICAL TRIAL: NCT01967199
Title: Treatment of Drug-Eluting Stent REstenosis Using Drug-Eluting STents vs. Drug-COated Balloon for Preventing REcurrent In-Stent Restenosis
Brief Title: Drug-eluting Stents vs. Drug-coated Balloon for Preventing Recurrent In-stent Restenosis
Acronym: RESTORE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, M.D, Ph.D., Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2013-01
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Coronary Restenosis
Keywords: drug-eluting stent; drug-coated Balloon; recurrent In-Stent restenosis
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Eluting Stent (Active Comparator): Everolimus-eluting balloon expandable stent (Xience Prime or Xience Xpedition or Xience Alpine)
  Interventions: Device: Everolimus-eluting balloon expandable stent
- paclitaxel eluting balloon (Experimental): paclitaxel eluting balloon (SeQuent Please)
  Interventions: Device: paclitaxel eluting balloon

INTERVENTIONS:
Device: Everolimus-eluting balloon expandable stent — Everolimus-eluting balloon expandable stent (Xience Prime or Xience Xpedition or Xience Alpine)
  Arms: Drug Eluting Stent
Device: paclitaxel eluting balloon — paclitaxel eluting balloon (SeQuent Please)
  Arms: paclitaxel eluting balloon

SUMMARY:
The purpose of this study is to establish the safety and effectiveness of paclitaxel eluting balloon (SeQuent Please) compared to coronary stenting with the Everolimus-eluting balloon expandable stent (Xience Prime or Xience Xpedition or Xience Alpine) in the treatment of drug eluting stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be more than or equal to 20 years of age
* Restenosis after drug-eluting stents (>50% by visual estimate)
* Any Lesion length including focal in stent restenosis or diffuse in stent restenosis
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications:

  * Heparin
  * Aspirin
  * Both Clopidogrel and TIclopidine
  * Sirolimus eluting stent
  * Stainless steel and/or
  * Contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled)
* Systemic (intravenous) Everolimus use within 12 months.
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2013-04-18 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Late luminal loss | 9months
  Late luminal loss at 9 months angiographic follow-up.

SECONDARY OUTCOMES:
Death | 1 year
Myocardial infarction | 1 year
Target lesion revascularization | 1 year
Target vessel revascularization | 1 year
Stent thrombosis | 1 year
In-segment or in-stent restenosis at 9 month angiographic follow-up | 1 year
Procedural success | 3day
  defined as achievement of a final diameter stenosis of <30% by QCA(Quantitative Coronary Angiography) using any percutaneous method, without the occurrence of death, Q wave Myocardial Infarction, or repeat revascularization of the target lesion during the hospital stay.
  participants will be followed for the duration of hospital stay, an expected average of 3days.

CONTACTS AND LOCATIONS:
Locations (11):
- South Korea (11):
  - Asan Medical Center, Seoul, Songpa-gu
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Chungbuk National University Hospital, Chungjoo
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - National Health Insurance Service Ilsan Hospital, Ilsan
  - Dong-A Medical Center, Pusan
  - Seoul National University Boramae Medical Center, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Wong YTA, Kang DY, Lee JB, Rha SW, Hong YJ, Shin ES, Her SH, Nam CW, Chung WY, Kim MH, Lee CH, Lee PH, Ahn JM, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Park DW, Park SJ. Comparison of drug-eluting stents and drug-coated balloon for the treatment of drug-eluting coronary stent restenosis: A randomized RESTORE trial. Am Heart J. 2018 Mar;197:35-42. doi: 10.1016/j.ahj.2017.11.008. Epub 2017 Nov 22. PMID 29447782